CLINICAL TRIAL: NCT05503082
Title: Ubrogepant Efficacy and Safety in the Treatment of Acute Migraine in Patients Currently Treated With CGRP Monoclonal Antibodies (CGRPmAbs)
Brief Title: Ubrogepant treatmeNt in mIgraine Patients Utilizing mOnoclonal aNtibodies
Acronym: UNION
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chicago Headache Center & Research Institute (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Bradley Torphy, MD, Managing Director, Chicago Headache Center & Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-02
Record Dates: First submitted 2022-08-14; First posted 2022-08-16 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Headache, Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — ubrogepant

STUDY DESIGN:
Intervention Model Description: Phase IV prospective open label randomized clinical study evaluating safety and efficacy of ubrogepant (UBRELVY) in patients currently treated with one of the injectable monoclonal antibodies targeting CGRP or the CGRP receptor (Aimovig, Ajovy, or Emgality).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- w/o CGRPmAb (Placebo Comparator): w/o CGRPmAb
  Interventions: Drug: Ubrogepant 50 MG [Ubrelvy]; Drug: Ubrogepant 100 MG [Ubrelvy]
- Tx w/ CGRPmAb (Active Comparator): Tx w/ CGRPmAb
  Interventions: Drug: Ubrogepant 50 MG [Ubrelvy]; Drug: Ubrogepant 100 MG [Ubrelvy]

INTERVENTIONS:
Drug: Ubrogepant 50 MG [Ubrelvy] — Ubrogepant 50 MG [Ubrelvy]
Drug: Ubrogepant 100 MG [Ubrelvy] — Ubrogepant 100 MG [Ubrelvy]

SUMMARY:
This is a prospective open-label randomized study assessing similar endpoints included in the pivotal trial for ubrogepant, which are pain freedom and freedom from the most bothersome symptom at two hours. Patients between 18-75 years old with a one-year history of migraine who experience ≥3 migraine days/month will be screened. This study will include migraine patients treated with or without injectable CGRPmAbs. As was the case in the clinical trials, this will be a single-attack study. Patients will be randomized to treat a single migraine attack with ubrogepant 50mg or 100mg. Patients will record dosing time, most bothersome symptom (nausea, photophobia, or phonophobia - chosen by patient), pain freedom, pain relief, the use of a 2nd dose if required, and adverse reactions. Patients will follow up within 30 days post treatment. Patients will be assessed for adverse events, and the safety data will be compared with the original clinical trial.

DETAILED DESCRIPTION:
The purpose of this study is to examine the safety and efficacy of ubrogepant (UBRELVY) in patients currently treated with one of the injectable monoclonal antibodies targeting CGRP or the CGRP receptor (Aimovig, Ajovy, or Emgality). There are currently very limited data available about the use of CGRP receptor antagonists in this population, resulting in difficulty obtaining prior authorization to use ubrogepant in patients currently treated with CGRPmAbs. Questions remain as to whether these patients, whose CGRP or CGRP receptors are suppressed, will experience the same safety and efficacy results as patients without such suppression by CGRPmAbs.

This is a prospective open-label randomized study assessing similar endpoints included in the pivotal trial for ubrogepant, which are pain freedom and freedom from the most bothersome symptom at two hours. Patients between 18-75 years old with a one-year history of migraine who experience ≥3 migraine days/month will be screened. This study will include migraine patients treated with or without injectable CGRPmAbs. As was the case in the clinical trials, this will be a single-attack study. Patients will be randomized to treat a single migraine attack with ubrogepant 50mg or 100mg. Patients will record dosing time, most bothersome symptom (nausea, photophobia, or phonophobia - chosen by patient), pain freedom, pain relief, the use of a 2nd dose if required, and adverse reactions. Patients will follow up within 30 days post treatment. Patients will be assessed for adverse events, and the safety data will be compared with the original clinical trial.

Primary Objective:

To evaluate the safety and efficacy of ubrogepant (UBRELVY) in patients currently treated with one of the injectable monoclonal antibodies targeting CGRP or the CGRP receptor (Aimovig, Ajovy, or Emgality).

Primary Endpoint:

* Pain freedom at 2 hours.
* Freedom from most bothersome symptom at 2 hours

Secondary Objectives:

To assess improvements with the addition of ubrogepant (UBRELVY) in patients currently treated with one of the injectable monoclonal antibodies targeting CGRP or the CGRP receptor (Aimovig, Ajovy, or Emgality).

Secondary Endpoint:

* Pain relief at 2 hours (this is different from pain freedom: moderate to severe pain reduced to mild or no pain)
* Percentage of patients with sustained pain relief from 2-24 hours after initial dose
* Percentage of patients with sustained pain freedom from 2-24 hours after initial dose
* Pain relief at 2 hours after 2nd dose
* Percentage of patients with sustained pain relief from 2-24 hours after 2nd dose
* Percentage of patients with sustained pain freedom from 2-24 hours after 2nd dose

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ages 18 to 75 years, at screening (Visit 1).
* At least a 1-year history of migraine with or without aura.
* History of ≥3 monthly headache days of at least moderate severity.
* Study patient currently on CGRPmAbs must be on treatment > 1 month at screening.
* By history, the patient's migraines typically last between 4 and 72 hours if untreated or treated unsuccessfully and migraine episodes are separated by at least 48 hours of headache pain freedom

Exclusion Criteria:

* History of <3 monthly headache days of at least moderate severity
* Concomitant use of strong CYP3A4 inducers (e.g., phenytoin, barbiturates, rifampin, St. John's Wort)
* Concomitant use of strong CYP3A4 inhibitors (e.g., ketoconazole, itraconazole, clarithromycin)
* Currently on Botox treatment for CM.
* Concomitant use of gepants as a preventative treatment.
* Current user of illicit drugs, or a history within 1 year prior to screening (visit 1) of drug or alcohol abuse or dependence
* Clinically significant hematologic, endocrine, cardiovascular, pulmonary, gastrointestinal, or neurologic disease. If there is a history of such a disease, but the condition has been stable for more than 1 year prior to screening (visit 1) and is judged by the PI as not likely to interfere with participation in the study, the participant may be included.
* Woman is pregnant, planning to become pregnant during the course of the study, or currently lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Pain freedom | 2 hours post treatment
  Pain freedom at 2 hours.
Freedom from most bothersome symptom | 2 hours post treatment
  Freedom from most bothersome symptom at 2 hours.

SECONDARY OUTCOMES:
Pain relief at 2 hours | 2 hours post treatment
  Pain relief at 2 hours (this is different from pain freedom: moderate to severe pain reduced to mild or no pain).
Percentage of patients with sustained pain relief from 2-24 hours after initial dose. | 2-24 hours after initial dose
  Percentage of patients with sustained pain relief from 2-24 hours after initial dose.
Percentage of patients with sustained pain freedom from 2-24 hours after initial dose. | 2-24 hours after initial dose
  Percentage of patients with sustained pain freedom from 2-24 hours after initial dose.
Pain relief at 2 hours after 2nd dose | 2 hours after 2nd dose
  Pain relief at 2 hours after 2nd dose.
Percentage of patients with sustained pain relief from 2-24 hours after 2nd dose. | 2-24 hours after 2nd dose
  Percentage of patients with sustained pain relief from 2-24 hours after 2nd dose.
Percentage of patients with sustained pain freedom from 2-24 hours after 2nd dose. | 2-24 hours after 2nd dose
  Percentage of patients with sustained pain freedom from 2-24 hours after 2nd dose.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Torphy, MD, Principal Investigator — Chicago Headache Center & Research Institute
Locations (2):
- United States (2):
  - Chicago Headache Center & Research Institute, Chicago, Illinois
  - Chicago Headache Center & Research Institute, Naperville, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dodick DW, Lipton RB, Ailani J, Halker Singh RB, Shewale AR, Zhao S, Trugman JM, Yu SY, Viswanathan HN. Ubrogepant, an Acute Treatment for Migraine, Improved Patient-Reported Functional Disability and Satisfaction in 2 Single-Attack Phase 3 Randomized Trials, ACHIEVE I and II. Headache. 2020 Apr;60(4):686-700. doi: 10.1111/head.13766. Epub 2020 Feb 19. PMID 32073660
- See also: Chicago Headache Center & Research Institute — https://chicagoheadache.com/clinical-trials/